CLINICAL TRIAL: NCT00414648
Title: Multicenter International Lymphangioleiomyomatosis Efficacy and Safety of Sirolimus Trial
Brief Title: Efficacy and Safety of Sirolimus in LAM
Acronym: MILES
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Cincinnati (Other)
Collaborators: Office of Rare Diseases (ORD) (NIH); FDA Office of Orphan Products Development (U.S. Federal Agency); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Principal Investigator, Francis McCormack, Professor, University of Cincinnati
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RDCRN 5702; U54RR019498-01 (NIH); FD-003362-01 (Other Grant/Funding Number: FDA Office of Orphan Product Development); NCT00408343 (obsolete NCT alias); NCT00720746 (obsolete NCT alias)
Record Dates: First submitted 2006-12-20; First posted 2006-12-21 (Estimated); Results first posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Lymphangioleiomyomatosis
Keywords: Lymphangiomyomatosis; mTOR
MeSH Terms: conditions — Lymphangioleiomyomatosis | interventions — Sirolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Unlabeled sirolimus tablets were provided by Pfizer. Identical appearing placebo tablets were obtained from a commercial source. Sirolimus levels were reported only to the medical monitor. To maintain the blind, when dose adjustments were made in the sirolimus group, a sham adjustment was also made in the placebo group
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes

ARMS (2):
- Active Agent (Sirolimus) (Experimental): Participants receive sirolimus daily for 1 year and are followed with serial pulmonary function tests, 6-minute walk tests, and symptom and QOL questionnaires over a 2-year period.
  Interventions: Drug: Sirolimus
- Placebo Arm (Placebo Comparator): Participants receive placebo daily for 1 year and followed with serial pulmonary function tests, 6-minute walk tests, and symptom and QOL questionnaires over a 2-year period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sirolimus — A sirolimus dose of 2 tablets (1 mg/tablet) per day for 1 year.
  Other Names: Rapamycin
  Arms: Active Agent (Sirolimus)
Drug: Placebo — A placebo dose of 2 tablets per day for 1 year.
  Other Names: Other names: placebo
  Arms: Placebo Arm

SUMMARY:
Lymphangioleiomyomatosis (LAM) is a rare lung disease of women that is caused by genetic mutations. It results in the uncontrolled growth of an unusual type of smooth muscle cell in the lung. These cells invade lung tissue, including the airways, blood vessels, and lymph vessels, and restrict the flow of air, blood, and lymph, respectively. Respiratory failure, lung collapse (pneumothorax), and pleural effusions (chylothorax) are hallmarks of the disease. This study will evaluate the safety and effectiveness of sirolimus, an inhibitor of the mTOR pathway, in stabilizing or improving lung function in people with LAM.

DETAILED DESCRIPTION:
LAM is an uncommon, progressive, cystic lung disease that predominantly affects young women. The disease is caused by mutations in tuberous sclerosis complex (TSC) genes, which regulate cellular pathways that control nutrient sensing, cell size, cell migration, and cell proliferation. Individuals with LAM often experience pneumothorax and chylothorax, as well progressive loss of lung function. Sirolimus is drug that was approved for the prevention of kidney transplant rejection. It directly affects the cellular pathway that causes LAM. This study will evaluate the safety and effectiveness of sirolimus in stabilizing or improving lung function in people with LAM.

Individuals interested in participating in this 2-year, double-blind study will first report to the study sites for pulmonary function testing to determine their eligibility for participation. Participants deemed eligible will be randomly assigned to receive either sirolimus or placebo for 1 year. Sirolimus or placebo will be administered in 2 tablet doses (2 mg for sirolimus) for the duration of the study. Study visits will occur at baseline, Week 3, every 3 months for 12 months, and months 18 and 24. Study visits will include a physical exam, questionnaires, a pregnancy test, blood and urine collection, and functional lung tests. A 6-minute walk test will occur at most study visits; a chest x-ray will be taken at baseline and month 24; and a volumetric computed tomography scan will occur at baseline, month 12, and month 24. Adverse events, medication side effects, and lung function will be assessed at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Signed and dated informed consent
* Diagnosis of LAM based on compatible chest CT scan and a) biopsy or cytology consistent with LAM, or b) presence of tuberous sclerosis, angiomyolipoma or chylous pleural effusion; or c) a VEGF-D level of at least 800 pg/ml
* Forced expiratory volume in one second (FEV1) of 70% or less of predicted value after administration of a bronchodilator

Exclusion Criteria:

* Known allergy to sirolimus
* History of heart attack, angina, or stroke due to clogging, narrowing, and hardening of the arteries and blood vessels
* Significant hematologic or hepatic abnormality (transaminase levels greater than three times the upper limit of normal, HCT less than 30%, platelets less than 80,000/cubic mm, adjusted absolute neutrophil count less than 1,000/cubic mm, total white blood cell count less than 3,000/cubic mm)
* Intercurrent infection at the time treatment with sirolimus begins
* Any surgery involving entry into a body cavity or requiring three or more sutures within 8 weeks of initiation of study drug
* Use of an investigational drug within the 30 days prior to random assignment
* Uncontrolled hyperlipidemia
* Previous lung transplant or currently on lung transplant list
* Unable to attend scheduled study visits
* Unable to perform pulmonary function tests
* Creatinine levels greater than 2.5 mg/dl
* Chylous ascites severe enough to affect diaphragmatic function
* Pleural effusion severe enough to affect pulmonary function, as determined by the study physician
* History of acute pneumothorax within the 2 months prior to study entry
* History of malignancy within the 2 years prior to study entry (except for squamous or basal cell skin cancer)
* Use of estrogen containing medication within the thirty days prior to randomization
* Unable or unwilling to use adequate contraception
* Pregnant, breastfeeding, or plans to become pregnant within the next 2 years

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 89 (Actual)
Dates: Start 2006-12; Primary Completion 2010-09 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francis X McCormack, MD, Principal Investigator — University of Cincinnati Medical Center Division of Pulmonary and Critical Care Medicine
Locations (13):
- United States (10):
  - University of California Los Angeles, Los Angeles, California
  - National Jewish Medical and Research Center, Denver, Colorado
  - University of Florida, Gainesville, Gainesville, Florida
  - National Heart, Lung, and Blood Institute, Bethesda, Maryland
  - Harvard's Brigham and Women's Hospital, Boston, Massachusetts
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Health Center at Tyler, Tyler, Texas
- Toronto General Hospital, Toronto, Ontario, Canada
- Japan (2):
  - National Kinki-Chou Hospital, Sakai, Osaka
  - Niigata University Medical and Dental Hospital, Niigata

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McCarthy C, Gupta N, Johnson SR, Yu JJ, McCormack FX. Lymphangioleiomyomatosis: pathogenesis, clinical features, diagnosis, and management. Lancet Respir Med. 2021 Nov;9(11):1313-1327. doi: 10.1016/S2213-2600(21)00228-9. Epub 2021 Aug 27. PMID 34461049
- [Background] Gupta N, Lee HS, Ryu JH, Taveira-DaSilva AM, Beck GJ, Lee JC, McCarthy K, Finlay GA, Brown KK, Ruoss SJ, Avila NA, Moss J, McCormack FX; NHLBI LAM Registry Group. The NHLBI LAM Registry: Prognostic Physiologic and Radiologic Biomarkers Emerge From a 15-Year Prospective Longitudinal Analysis. Chest. 2019 Feb;155(2):288-296. doi: 10.1016/j.chest.2018.06.016. Epub 2018 Jun 22. PMID 29940164
- [Background] Ryu JH, Moss J, Beck GJ, Lee JC, Brown KK, Chapman JT, Finlay GA, Olson EJ, Ruoss SJ, Maurer JR, Raffin TA, Peavy HH, McCarthy K, Taveira-Dasilva A, McCormack FX, Avila NA, Decastro RM, Jacobs SS, Stylianou M, Fanburg BL; NHLBI LAM Registry Group. The NHLBI lymphangioleiomyomatosis registry: characteristics of 230 patients at enrollment. Am J Respir Crit Care Med. 2006 Jan 1;173(1):105-11. doi: 10.1164/rccm.200409-1298OC. Epub 2005 Oct 6. PMID 16210669
- [Background] Gupta N, Finlay GA, Kotloff RM, Strange C, Wilson KC, Young LR, Taveira-DaSilva AM, Johnson SR, Cottin V, Sahn SA, Ryu JH, Seyama K, Inoue Y, Downey GP, Han MK, Colby TV, Wikenheiser-Brokamp KA, Meyer CA, Smith K, Moss J, McCormack FX; ATS Assembly on Clinical Problems. Lymphangioleiomyomatosis Diagnosis and Management: High-Resolution Chest Computed Tomography, Transbronchial Lung Biopsy, and Pleural Disease Management. An Official American Thoracic Society/Japanese Respiratory Society Clinical Practice Guideline. Am J Respir Crit Care Med. 2017 Nov 15;196(10):1337-1348. doi: 10.1164/rccm.201709-1965ST. PMID 29140122
- [Background] McCormack FX, Gupta N, Finlay GR, Young LR, Taveira-DaSilva AM, Glasgow CG, Steagall WK, Johnson SR, Sahn SA, Ryu JH, Strange C, Seyama K, Sullivan EJ, Kotloff RM, Downey GP, Chapman JT, Han MK, D'Armiento JM, Inoue Y, Henske EP, Bissler JJ, Colby TV, Kinder BW, Wikenheiser-Brokamp KA, Brown KK, Cordier JF, Meyer C, Cottin V, Brozek JL, Smith K, Wilson KC, Moss J; ATS/JRS Committee on Lymphangioleiomyomatosis. Official American Thoracic Society/Japanese Respiratory Society Clinical Practice Guidelines: Lymphangioleiomyomatosis Diagnosis and Management. Am J Respir Crit Care Med. 2016 Sep 15;194(6):748-61. doi: 10.1164/rccm.201607-1384ST. PMID 27628078
- [Result] McCormack FX, Inoue Y, Moss J, Singer LG, Strange C, Nakata K, Barker AF, Chapman JT, Brantly ML, Stocks JM, Brown KK, Lynch JP 3rd, Goldberg HJ, Young LR, Kinder BW, Downey GP, Sullivan EJ, Colby TV, McKay RT, Cohen MM, Korbee L, Taveira-DaSilva AM, Lee HS, Krischer JP, Trapnell BC; National Institutes of Health Rare Lung Diseases Consortium; MILES Trial Group. Efficacy and safety of sirolimus in lymphangioleiomyomatosis. N Engl J Med. 2011 Apr 28;364(17):1595-606. doi: 10.1056/NEJMoa1100391. Epub 2011 Mar 16. PMID 21410393
- [Result] Argula RG, Kokosi M, Lo P, Kim HJ, Ravenel JG, Meyer C, Goldin J, Lee HS, Strange C, McCormack FX; MILES Study Investigators. A Novel Quantitative Computed Tomographic Analysis Suggests How Sirolimus Stabilizes Progressive Air Trapping in Lymphangioleiomyomatosis. Ann Am Thorac Soc. 2016 Mar;13(3):342-9. doi: 10.1513/AnnalsATS.201509-631OC. PMID 26799509
- [Result] Gupta N, Lee HS, Young LR, Strange C, Moss J, Singer LG, Nakata K, Barker AF, Chapman JT, Brantly ML, Stocks JM, Brown KK, Lynch JP 3rd, Goldberg HJ, Downey GP, Taveira-DaSilva AM, Krischer JP, Setchell K, Trapnell BC, Inoue Y, McCormack FX; NIH Rare Lung Disease Consortium. Analysis of the MILES cohort reveals determinants of disease progression and treatment response in lymphangioleiomyomatosis. Eur Respir J. 2019 Apr 4;53(4):1802066. doi: 10.1183/13993003.02066-2018. Print 2019 Apr. PMID 30846465
- [Result] Young L, Lee HS, Inoue Y, Moss J, Singer LG, Strange C, Nakata K, Barker AF, Chapman JT, Brantly ML, Stocks JM, Brown KK, Lynch JP 3rd, Goldberg HJ, Downey GP, Swigris JJ, Taveira-DaSilva AM, Krischer JP, Trapnell BC, McCormack FX; MILES Trial Group. Serum VEGF-D a concentration as a biomarker of lymphangioleiomyomatosis severity and treatment response: a prospective analysis of the Multicenter International Lymphangioleiomyomatosis Efficacy of Sirolimus (MILES) trial. Lancet Respir Med. 2013 Aug;1(6):445-52. doi: 10.1016/S2213-2600(13)70090-0. PMID 24159565
- [Result] Lo P, Brown MS, Kim H, Kim H, Argula R, Strange C, Goldin JG. Cyst-based measurements for assessing lymphangioleiomyomatosis in computed tomography. Med Phys. 2015 May;42(5):2287-95. doi: 10.1118/1.4916655. PMID 25979023
- [Derived] Harun N, Gupta N, McCormack FX, Macaluso M. Dynamic use of historical controls in clinical trials for rare disease research: A re-evaluation of the MILES trial. Clin Trials. 2023 Jun;20(3):223-234. doi: 10.1177/17407745231158906. Epub 2023 Mar 17. PMID 36927115
- [Derived] Xu KF, Wang L, Tian XL, Gui YS, Peng M, Cai BQ, Zhu YJ. The St. George's Respiratory Questionnaire in lymphangioleiomyomatosis. Chin Med Sci J. 2010 Sep;25(3):140-5. doi: 10.1016/s1001-9294(10)60038-7. PMID 21180274
- See also: Click here for the Health Informatics Institute of the University of South Florida — https://dm.hiidatacenter.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in December, 2006 and ended in August 2009. Recruitment occurred at the hospital based study sites.
Groups:
- Sirolimus Treatment Arm: Participants will receive sirolimus daily for 1 year followed with serial pulmonary functional tests and 6-minute walk tests over a 2-year period. Note: study truncated to 1 year with daily sirolimus in 2010. Second year of follow up eliminated after August 31, 2010.
- Placebo Treatment Arm: Participants will receive placebo sirolimus daily for 1 year followed with serial pulmonary functional tests and 6-minute walk tests over a 2-year period. Note: study truncated to 1 year with daily placebo sirolimus in 2010. Second year of follow up eliminated after August 31, 2010.
Period: Overall Study
Arm/Group | Sirolimus Treatment Arm | Placebo Treatment Arm
Started | 46 (46 participants were randomized to the sirolimus treatment arm.) | 43 (43 participants were randomized to the placebo treatment arm.)
Completed | 41 (41 participants in the sirolimus treatment arm had 12 month data available for analysis.) | 34 (34 participants in the placebo treatment arm had 12 month data available for analysis.)
Not Completed | 5 | 9
Not completed — Adverse Event | 5 | 5
Not completed — Death | 0 | 1
Not completed — Lack of Efficacy | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sirolimus Treatment Arm | Placebo Treatment Arm | Total
Number analyzed (Participants) | 46 | 43 | 89
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 46 | 43 | 89
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 43 | 89
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 15 | 12 | 27
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 29 | 30 | 59
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Changes in Forced Expiratory Volume in One-second (FEV1) Slope in Milliliters Per Month
Description: FEV1 values reported are in liters or milliliters. There are no definite minimum and maximum values of FEV1 as it is a physiological measure of lung function and varies from individual to individual. Normative ranges are determined in populations stratified by gender, height, age and race/ethnicity. Higher FEV1 values indicate better lung function.
Time Frame: Baseline to Month 12
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: milliliters per month
Groups:
- Sirolimus: sirolimus treatment arm FEV1 at 12 months.
- Placebo: Placebo arm FEV1 at 12 months
Arm/Group | Sirolimus | Placebo
Number analyzed (Participants) | 46 | 43
milliliters per month | 1 (2) | -12 (2)
Statistical Analysis 1: Comparison: Sirolimus vs Placebo; FEV1 slope; Test type: Superiority or Other; p < 0.001, Regression, Linear — The model included the time since enrollment, the treatment assignment, and the interaction between time and treatment; Mixed model with the use of the Kenward-Roger correction without imputation of missing data

2. Secondary Outcome: Percent of Participants With Serious Adverse Events
Time Frame: Baseline to Month 12
Population: Intention to treat
Measure: Number; unit: percentage of participants with SAE
Groups:
- Active Agent (Sirolimus): Participants received sirolimus daily for 1 year and were followed with serial pulmonary function tests and 6-minute walk tests over a 2-year period.
  Sirolimus: Initial sirolimus dose of 2 mg was given in the form of 2 tablets (1 mg/tablet) per day for 1 year, and was titrate to maintain a serum level of 5-10 ng/ml.
- Placebo Arm: Participants receive placebo daily for 1 year and were followed with serial pulmonary function tests and 6-minute walk tests over a 2-year period.
  Placebo sirolimus: Placebo was administered as 2 tablets per day for 1 year, and was sham adjusted in some subjects to maintain the blind.
Arm/Group | Active Agent (Sirolimus) | Placebo Arm
Number analyzed (Participants) | 46 | 43
percentage of participants with SAE | 50 | 41.86
Statistical Analysis 1: Comparison: Active Agent (Sirolimus) vs Placebo Arm; Test type: Other; p = .441, Chi-squared

3. Secondary Outcome: Changes in FVC Slope in ml/Month
Description: FVC values are reported in liters or milliliters. Normative ranges are determined in populations that are stratified by gender, height, age and race/ethnicity. There are no minimum or maximum values as it is a physiologic measure of lung function and varies from individual to individual. Higher FVC scores indicate better lung function.
Time Frame: Baseline to Month 12
Population: Intention To Treat
Measure: Mean (Standard Deviation); unit: milliliters/month
Groups:
- Sirolimus Treatment Arm: Participants received sirolimus daily for 1 year and were followed with serial pulmonary function tests and 6-minute walk tests over a 2-year period.
- Placebo Treatment Arm: Participants received placebo daily for 1 year followed with serial pulmonary function tests and 6-minute walk tests over a 2-year period.
Arm/Group | Sirolimus Treatment Arm | Placebo Treatment Arm
Number analyzed (Participants) | 46 | 43
milliliters/month | 8 (3) | -11 (3)
Statistical Analysis 1: Comparison: Sirolimus Treatment Arm vs Placebo Treatment Arm; Test type: Superiority or Other; p = 0.001, Regression, Linear; GLM adjusted for baseline

4. Secondary Outcome: Rate of Change in Diffusing Capacity for Carbon Monoxide (DLCO) in ml/Min/mmHg
Description: Diffusing capacity for carbon monoxide is abbreviated DLCO. DLCO is measured in liters and milliliters. There are no definite minimum and maximum values of FEV1 as it is a physiological measure of lung function and varies from individual to individual. A lower DLCO means that there is lower lung function.
Time Frame: Baseline to Month 12
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: ml/min/mmHg
Arm/Group | Sirolimus Treatment Arm | Placebo Treatment Arm
Number analyzed (Participants) | 46 | 43
ml/min/mmHg | -0.01 (0.02) | -0.06 (0.03)
Statistical Analysis 1: Comparison: Sirolimus Treatment Arm vs Placebo Treatment Arm; Test type: Superiority or Other; p = 0.17, Regression, Linear; GLM adjusted for baseline

5. Secondary Outcome: Rate of Change in Total Lung Volume in ml Per Month
Description: There are two methods for measurement of total lung volume, nitrogen or helium wash out (total lung capacity or TLC), or plethysmography (Total gas volume or TGV). TLC or TGV is measured in milliliters or liters. Normative ranges for TLC or TGV are stratified by age, height, and sex in population based studies of normal subjects.. There are no definite minimum and maximum values of lung volume as it is a physiological measure of lung function and varies from individual to individual. A low TGV or TLC is suggestive of a restrictive lung disease, and a high TGV or TLC is consistent with obstructive lung disease with hyperinflation.
Time Frame: Baseline to Month 12
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: milliliters/month
Arm/Group | Sirolimus Treatment Arm | Placebo Treatment Arm
Number analyzed (Participants) | 46 | 43
milliliters/month | 8 (7) | -2 (7)
Statistical Analysis 1: Comparison: Sirolimus Treatment Arm vs Placebo Treatment Arm; Test type: Superiority; p = 0.34, Regression, Linear; GLM adjusted for baseline

6. Secondary Outcome: Rate of Change in Six Minute Walk Distance in Meters/Month
Description: Number of meters walked in six minutes. There is no minimum or maximum number of feet walked as this varies from individual to individual. A higher number of feet walked indicates better exercise tolerance
Time Frame: Baseline to Month 12
Population: Intention to treat
Measure: Mean (Standard Deviation); unit: meters/month
Groups:
- Sirolimus Treatment Arm: Participants received sirolimus daily for 1 year followed with serial pulmonary function tests and 6-minute walk tests over a 2-year period.
Arm/Group | Sirolimus Treatment Arm | Placebo Treatment Arm
Number analyzed (Participants) | 46 | 43
meters/month | 1.65 (0.81) | 1.47 (0.87)
Statistical Analysis 1: Comparison: Sirolimus Treatment Arm vs Placebo Treatment Arm; Test type: Superiority or Other; p = 0.88, Regression, Linear; GLM adjusted for baseline

7. Secondary Outcome: Rate of Change in Serum Vascular Endothelial Growth Factor-D (VEGF-D) Levels in pg/ml Per Month
Description: Serum VEGF-D is a protein produced by LAM cells that serves as a biomarker of mTOR activation and sirolimus response. Mean serum levels of VEGF-D in normal subjects are around 350 pg/ml. Higher levels of serum VEGF-D are correlated with greater degrees of mTOR activation, and a fall in VEGF-D levels suggest suppression of the mTOR axis.
Time Frame: Baseline to Month 12
Measure: Mean (Standard Deviation); unit: pg/ml per month
Groups:
- Placebo Treatment Arm: Participants received placebo daily for 1 year and were followed with serial pulmonary function tests and 6-minute walk tests over a 2-year period.
Arm/Group | Sirolimus Treatment Arm | Placebo Treatment Arm
Number analyzed (Participants) | 46 | 43
pg/ml per month | -88.01 (16.61) | -2.42 (17.23)
Statistical Analysis 1: Comparison: Sirolimus Treatment Arm vs Placebo Treatment Arm; Test type: Superiority or Other; p = 0.001, Regression, Linear; GLM adjusted for baseline

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over a 2 year period (12 month treatment period and 12 month observation period).
Arm/Group | Sirolimus Treatment Arm | Placebo Treatment Arm
All-Cause Mortality (participants affected / at risk) | 0/46 | 1/43
Serious Adverse Events (participants affected / at risk) | 23/46 | 18/43
Other Adverse Events (participants affected / at risk) | 46/46 | 43/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sirolimus Treatment Arm (N=46) | Placebo Treatment Arm (N=43)
Cardiac (Cardiac disorders) | 1 (1) | 0 (0)
blood or bone marrow (Blood and lymphatic system disorders) | 5 (5) | 0 (0)
Gastrointestinal (Gastrointestinal disorders) | 3 (3) | 1 (1)
Infection (Infections and infestations) | 2 (2) | 3 (3)
Metabolic (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 7 (7) | 1 (1)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 13 (13)
Vascular (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sirolimus Treatment Arm (N=46) | Placebo Treatment Arm (N=43)
"Blood and lymphatic system disorders - Other, specify" (Blood and lymphatic system disorders) | 2 (2) | 2 (4)
Anemia (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
"Blood and lymphatic system disorders - Other, specify" (Blood and lymphatic system disorders) | 1 (1) | 4 (7)
"Cardiac disorders - Other, specify" (Cardiac disorders) | 4 (7) | 4 (5)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 1 (2)
Pericardial effusion (Cardiac disorders) | 3 (4) | 2 (2)
Supraventricular tachycardia (Cardiac disorders) | 2 (4) | 0 (0)
"Ear and labyrinth disorders - Other, specify" (Ear and labyrinth disorders) | 1 (1) | 1 (1)
External ear inflammation (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Middle ear inflammation (Ear and labyrinth disorders) | 3 (3) | 1 (1)
External ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1)
"Endocrine disorders - Other, specify" (Endocrine disorders) | 2 (2) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 2 (2) | 0 (0)
Conjunctivitis (Eye disorders) | 1 (1) | 0 (0)
"Eye disorders - Other, specify" (Eye disorders) | 5 (7) | 3 (3)
Flashing lights (Eye disorders) | 0 (0) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 1 (2) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3) | 1 (1)
Periodontal disease (Gastrointestinal disorders) | 1 (4) | 1 (1)
Dental caries (Gastrointestinal disorders) | 2 (6) | 3 (3)
Diarrhea (Gastrointestinal disorders) | 29 (80) | 14 (54)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 2 (3) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (2)
Flatulence (Gastrointestinal disorders) | 2 (4) | 0 (0)
Gastritis (Gastrointestinal disorders) | 2 (2) | 1 (1)
"Gastrointestinal disorders - Other, specify" (Gastrointestinal disorders) | 13 (19) | 13 (17)
Dyspepsia (Gastrointestinal disorders) | 5 (5) | 4 (16)
Hemorrhoids (Gastrointestinal disorders) | 3 (4) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 16 (53) | 9 (17)
Mucositis oral (Gastrointestinal disorders) | 25 (67) | 22 (48)
Nausea (Gastrointestinal disorders) | 18 (31) | 11 (17)
Abdominal pain (Gastrointestinal disorders) | 6 (9) | 1 (2)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 5 (8) | 5 (6)
"General disorders and administration site conditions - Other, specify" (General disorders) | 1 (1) | 3 (5)
Sudden death NOS (General disorders) | 0 (0) | 1 (1)
Edema face (General disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 11 (13) | 7 (7)
Fatigue (General disorders) | 14 (21) | 13 (20)
Fever (General disorders) | 6 (8) | 4 (4)
Pain (General disorders) | 24 (63) | 20 (48)
Non-cardiac chest pain (General disorders) | 10 (12) | 7 (12)
Chills (General disorders) | 4 (5) | 3 (3)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
"Hepatobiliary disorders - Other, specify" (Hepatobiliary disorders) | 0 (0) | 1 (1)
Allergic reaction (Immune system disorders) | 0 (0) | 2 (2)
"Immune system disorders - Other, specify" (Immune system disorders) | 4 (6) | 3 (3)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0)
"Infections and infestations - Other, specify" (Infections and infestations) | 0 (0) | 1 (1)
"Infections and infestations - Other, specify" (Infections and infestations) | 32 (98) | 24 (79)
Bronchial infection (Infections and infestations) | 0 (0) | 1 (5)
Lung infection (Infections and infestations) | 0 (0) | 1 (1)
Mucosal infection (Infections and infestations) | 0 (0) | 1 (1)
Gum infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 0 (0) | 2 (2)
Upper respiratory infection (Infections and infestations) | 2 (2) | 2 (2)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 5 (10) | 4 (6)
Burn (Injury, poisoning and procedural complications) | 1 (1) | 2 (3)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Postoperative thoracic procedure complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 4 (4) | 1 (2)
Aspartate aminotransferase increased (Investigations) | 6 (7) | 3 (6)
Alkaline phosphatase increased (Investigations) | 2 (2) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Cholesterol high (Investigations) | 9 (11) | 6 (6)
Creatinine increased (Investigations) | 0 (0) | 1 (1)
Forced expiratory volume decreased (Investigations) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 4 (4) | 0 (0)
Lymphocyte count decreased (Investigations) | 3 (3) | 0 (0)
"Investigations - Other, specify" (Investigations) | 13 (20) | 2 (2)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0)
Weight gain (Investigations) | 0 (0) | 1 (1)
Weight loss (Investigations) | 5 (7) | 2 (2)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 3 (3) | 2 (3)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (3) | 2 (3)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Glucose intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 4 (4) | 2 (4)
Hyperuricemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Joint range of motion decreased cervical spine (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 2 (4) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Joint range of motion decreased lumbar spine (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
"Musculoskeletal and connective tissue disorder - Other, specify" (Musculoskeletal and connective tissue disorders) | 18 (28) | 12 (19)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 5 (6)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 3 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (5)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (6) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 9 (21) | 9 (13)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Memory impairment (Nervous system disorders) | 1 (2) | 1 (1)
"Nervous system disorders - Other, specify" (Nervous system disorders) | 5 (6) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 2 (4)
Headache (Nervous system disorders) | 13 (33) | 12 (27)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Sinus pain (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0)
Dysgeusia (Nervous system disorders) | 1 (1) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 7 (7) | 5 (5)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 3 (3) | 3 (4)
Depression (Psychiatric disorders) | 4 (4) | 4 (4)
Psychosis (Psychiatric disorders) | 0 (0) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 2 (3) | 2 (3)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 3 (3) | 1 (1)
"Renal and urinary disorders - Other, specify" (Renal and urinary disorders) | 5 (6) | 3 (4)
Urinary frequency (Renal and urinary disorders) | 3 (3) | 1 (1)
Uterine hemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Irregular menstruation (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine pain (Reproductive system and breast disorders) | 0 (0) | 1 (3)
"Reproductive system and breast disorders - Other, specify" (Reproductive system and breast disorders) | 2 (2) | 4 (5)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal dryness (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Vaginal inflammation (Reproductive system and breast disorders) | 0 (0) | 2 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 3 (9)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 5 (5)
Cough (Respiratory, thoracic and mediastinal disorders) | 18 (28) | 16 (25)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 12 (18) | 17 (34)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 (6) | 2 (6)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (3)
Laryngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 4 (7) | 4 (6)
Pharyngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (3)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 4 (5)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 6 (11)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
"Respiratory, thoracic and mediastinal disorders - Other, specify" (Respiratory, thoracic and mediastinal disorders) | 27 (55) | 26 (49)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
"Skin and subcutaneous tissue disorders - Other, specify" (Skin and subcutaneous tissue disorders) | 19 (30) | 8 (15)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0)
Skin induration (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nail loss (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Photosensitivity (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 5 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 (11) | 7 (8)
Rash acneiform (Skin and subcutaneous tissue disorders) | 20 (50) | 5 (6)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 (4) | 2 (2)
Telangiectasia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin ulceration (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
"Vascular disorders - Other, specify" (Vascular disorders) | 5 (6) | 3 (5)
Hot flashes (Vascular disorders) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 4 (4) | 5 (5)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0)
"Vascular disorders - Other, specify" (Vascular disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
The observation period of the trial was truncated for some subjects, driven by funding limitations, need for timely reporting and drug expiration factors. Please see supplement to McCormack FX, et al. Efficacy and safety of sirolimus in LAM. N Engl J Med. 2011, 28;364:1595-606. PMID: 21410393 for more detail.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No